CLINICAL TRIAL: NCT05429372
Title: A PHASE 2, MULTICENTER, SINGLE-ARM STUDY TO EVALUATE THE SAFETY AND DYSTROPHIN EXPRESSION AFTER FORDADISTROGENE MOVAPARVOVEC (PF-06939926) ADMINISTRATION IN MALE PARTICIPANTS WITH EARLY STAGE DUCHENNE MUSCULAR DYSTROPHY
Brief Title: Study of Fordadistrogene Movaparvovec in Early Stage Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: All participants who have received fordadistrogene movaparvovec in any Pfizer study will now be assessed for long-term safety in one combined study: C3391003
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3391008; 2021-003379-33 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2022-06-23 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Early Stage Duchenne Muscular Dystrophy; DMD; gene therapy; fordadistrogene movaparvovec
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06939926 (Experimental)
  Interventions: Genetic: PF-06939926

INTERVENTIONS:
Genetic: PF-06939926 — All participants will receive a single dose of PF-06939926 on Day 1.
  Other Names: Fordadistrogene Movaparvovec

SUMMARY:
The study will evaluate the safety and dystrophin expression following gene therapy in boys with Duchenne Muscular Dystrophy (DMD). It is a single-arm, non-randomized, open-label study

DETAILED DESCRIPTION:
The study will assess the safety and tolerability of fordadistrogene movaparvovec gene therapy. Approximately 10 participants will be enrolled in the study and receive a single IV infusion of PF-06939926; there is no placebo arm. The study includes boys who are at least 2 years old and less than 4 years old (including 3 year olds up until their 4th birthday). All boys will need to be negative for neutralizing antibodies against AAV9, as measured by the test done for the study as part of screening.

The primary analysis will occur when all participants have completed visits through Week 52 (or withdrawn from the study prior to Week 52). All participants will be followed in the study for 5 years after treatment with gene therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DMD by prior genetic testing.

Exclusion Criteria:

* Any of the following genetic abnormalities in the dystrophin gene: a. Any mutation (exon deletion, exon duplication, insertion, or point mutation) affecting any exon between exon 9 and exon 13, inclusive; OR b. A deletion that affects both exon 29 and exon 30; OR c. A deletion that affects any exons between 56-71, inclusive.
* Positive test performed by Pfizer for neutralizing antibodies to AAV9.
* Any prior treatment with gene therapy.
* Any treatment designed to increase dystrophin expression within 6 months prior to screening (including, but not limited to, exon-skipping and nonsense read through).
* Previous or current treatment with oral glucocorticoids or other immunosuppressive agents for the indication of DMD.
* Abnormality in specified laboratory tests, including blood counts, liver and kidney function.

Ages: 2 Years to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male participants age ≥2 to <4 years, at Screening (Visit 1)
Enrollment: 10 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events and Serious Adverse Events | Through Week 52
Number of participants with abnormal hematology test results | Through Week 52
  Blood samples will be collected from subjects for the analysis of hematology
Number of participants with abnormal biochemistry test results | Through Week 52
  Blood samples will be collected from subjects for the analysis of biochemistry
Number of participants with abnormal urine analysis | Through Week 52
  Urine samples will be collected from subjects for the analysis of urine
Number of participants with abnormal and clinically relevant changes in neurological examinations | Through Week 52
Number of participants with abnormal and clinically relevant changes in body weight | Through Week 52
Number of participants with abnormal and clinically relevant changes in vital signs | Through Week 52
Number of participants with abnormal and clinically relevant changes on cardiac troponin I | Through Week 52
Number of participants with abnormal and clinically relevant changes on electrocardiogram (ECG) | Through Week 52
Number of participants with abnormal and clinically relevant changes on echocardiogram | Through Week 52

SECONDARY OUTCOMES:
Distribution of mini-dystrophin expression in muscle | At Week 9, Week 52 and Year 5 (if available)
  Mini-dystrophin distribution from a muscle biopsy will be assessed by immunofluorescence
Level of mini-dystrophin expression in muscle | At Week 9, Week 52 and Year 5 (if available)
  Mini-dystrophin expression level from a muscle biopsy will be assessed by liquid chromatography mass spectrometry
Incidence and severity of Treatment-Emergent Adverse Events and Serious Adverse Events | Through 5 years
Number of participants with abnormal hematology test results | Through 5 years
  Blood samples will be collected from subjects for the analysis of hematology
Number of participants with abnormal biochemistry test results | Through 5 years
  Blood samples will be collected from subjects for the analysis of biochemistry
Number of participants with abnormal urine analysis | Through 5 years
  Urine samples will be collected from subjects for the analysis of urine
Number of participants with abnormal and clinically relevant changes in neurological examinations | Through 5 years
Number of participants with abnormal and clinically relevant changes in body weight | Through 5 years
Number of participants with abnormal and clinically relevant changes in vital signs | Through 5 years
Number of participants with abnormal and clinically relevant changes on cardiac troponin I | Through 5 years
Number of participants with abnormal and clinically relevant changes on electrocardiogram (ECG) | Through 5 years
Number of participants with abnormal and clinically relevant changes on echocardiogram | Through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (9):
  - UF Health Shands Hospital, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - CTSI Clinical Research Center, Salt Lake City, Utah
  - University of Utah Imaging and Neurosciences Center, Salt Lake City, Utah
  - University of Utah Hospital & Clinics Investigational Drug Services, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - The Royal Children's Hospital Melbourne, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3391008